CLINICAL TRIAL: NCT00879242
Title: Multicenter, Open Label, Prospective Study to Evaluate the Efficacy and Safety of Deferasirox 30 mg/kg/Day for 52 Weeks, in Transfusion-dependent Beta-thalassemic Patients With Cardiac MRI T2* < 20 Msec
Brief Title: Effect of Deferasirox on Patients With Cardiac MRI T2* < 20 Msec
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CICL670AIT07; EUDRACT Code :2008-003230-22
Record Dates: First submitted 2009-04-08; First posted 2009-04-09 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2011-11

CONDITIONS: Beta Thalassemia Transfusion Dependent
Keywords: Thalassemia; cardiac MRI T2*
MeSH Terms: conditions — Thalassemia | interventions — Deferasirox

ARMS (1):
- Deferasirox (Experimental): 30 mg/kg/day. The daily dose can be increased to 40 mg/kg in case of unsatisfactory response after 12 weeks of treatment.
  Interventions: Drug: Deferasirox

INTERVENTIONS:
Drug: Deferasirox — Dispersible tables of 125, 250 and 500 mg at the dose of 30 mg/kg/day, oral administration.

SUMMARY:
This study will assess the safety and efficacy of deferasirox in patients with cardiac MRI T2* < 20 msec.

ELIGIBILITY:
Inclusion Criteria:

* β-thalassemic patients receiving regular transfusions with an history of at least 20 transfusional events
* Patients naïve for deferasirox
* Serum ferritin levels ≥1000ng/ml (average of the last 6 months assays);
* Cardiac MRI T2* >5 and <20 msec.
* LVEF at MRI ≥56%

Exclusion Criteria:

* Patients that have already started deferasirox therapy
* Existing contraindications to the performance of MRI procedure, including presence of metallic prostheses not compatible with the MRI procedure other than those approved as safe for use in MRI scanners (e.g., some types of aneurysm clips, shrapnel in proximity to vital organs such as the retina), pacemaker, intractable claustrophobia and incapability to follow the instruction for the correct performance of the MRI (e.g. to maintain a supine position, to hold breath, etc.)
* Clinical conditions requiring intensive chelating therapy on the basis of Investigator's judgment
* Stable average ALT levels >300 U/L in the preceding 12 months
* Uncontrolled systemic hypertension
* Estimated creatinine clearance <60 ml/min
* History of nephrotic syndrome
* History of clinically significant ocular toxicity related to the chelating therapy
* Psychiatric disorders or drug dependence that might impair the capability of the patient to provide their Informed Consent or to be administered the study treatment
* Known sensitivity to study drug(s) or class of study drug(s)
* Patients with severe medical condition(s) that in the view of the investigator prohibits participation in the study
* Use of any other investigational agent in the last 30 days.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-02; Primary Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in cardiac T2* value | 52 weeks
  Unsatisfactory response is a monthly MRI T2* improvement lower than 3% versus baseline.

SECONDARY OUTCOMES:
Change from baseline in cardiac functions parameters (LVEF, LVESV and LVEDV) | 52 weeks
Change from baseline liver T2* value | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Italy (2):
  - Novartis Investigative Site, Cagliari
  - Novartis Investigative Site, Orbassano

REFERENCES:
- [Result] Piga A, Longo F, Origa R, Roggero S, Pinna F, Zappu A, Castiglioni C, Cappellini MD. Deferasirox for cardiac siderosis in beta-thalassaemia major: a multicentre, open label, prospective study. Br J Haematol. 2014 Nov;167(3):423-6. doi: 10.1111/bjh.12987. Epub 2014 Jun 30. No abstract available. PMID 24976388